CLINICAL TRIAL: NCT05336760
Title: Dysphagia, Quality of Life and Attitudes Towards Percutaneous Endoscopic Gastrostomy in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Dysphagia, QoL and Attitudes Towards PEG in ALS Patients
Acronym: ALSDPEG
Status: Recruiting | Type: Observational
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: URIS202201
Record Dates: First submitted 2022-03-16; First posted 2022-04-20 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALS Patients: Patients with confirmed amyotrophic lateral sclerosis.
  Interventions: Diagnostic Test: Iowa Oral Performance Instrument (IOPI); Diagnostic Test: Mann Assessment of Swallowing Ability (MASA); Diagnostic Test: Fiberoptic Endoscopic Evaluation of Swallowing; Diagnostic Test: Respiratory function measurements
- Relatives: Close relatives of the patients included in the study.

INTERVENTIONS:
Diagnostic Test: Iowa Oral Performance Instrument (IOPI) — IOPI measures the peak pressure of the tongue strength and endurance using a disposable bulb placed on a hard palate behind the front teeth or at the base of the tongue. The participants will be asked to press the bulb with their tongue with maximum pressure, three times. To measure the endurance, the participants will be asked to hold the pressure for as long as they can.
  Groups: ALS Patients
Diagnostic Test: Mann Assessment of Swallowing Ability (MASA) — MASA is a standard clinical swallowing assessment protocol including general patient examination, on-the-outside visible signs of oral preparatory and transportation phase and pharyngeal phase of swallowing function.
  Groups: ALS Patients
Diagnostic Test: Fiberoptic Endoscopic Evaluation of Swallowing — The subjects will ingest up to 10 boluses ranging in thickness and volume (from thin to extremely-thick and a cookie).
  Groups: ALS Patients
Diagnostic Test: Respiratory function measurements — Respiratory function measurements will include forced vital capacity (FVC), maximum inspiratory pressure (MIP), and maximum expiratory pressure (MEP), all expressed in percentage of predicted values. Conventional methods of testing will be applied.
  Groups: ALS Patients

SUMMARY:
In Amyotrophic Lateral Sclerosis, dysphagia has a high incidence. With deterioration of swallowing function, percutaneous endoscopic gastrostomy (PEG) tube is recommended to ensure sufficient and safe oral intake. Dysphagia and PEG placement alter quality of life (QoL). However, QoL and attitudes toward PEG remain largely unexplored. The purpose of this study is to monitor the swallowing function in relationship to QoL and attitudes toward PEG tube insertion and feeding.

DETAILED DESCRIPTION:
The purpose of this study is to monitor the deterioration of swallowing function in ALS patient population, and to explore its impact on QoL and attitudes toward PEG tube insertion and feeding in the course of the disease. It will take maximum of 60 minutes to fully evaluate the swallowing function and complete the questionnaires. The evaluation procedure will be repeated every 3 months until PEG tube insertion, which will allow us to closely monitor the swallowing function in a relation to attitudes toward PEG and QoL. The data obtained from this study should contribute significantly to the knowledge of QoL in ALS patients with dysphagia, and it will allow for a comparison of QoL in ALS patients with and without PEG tube. This study will also expand the understanding of attitudes in ALS patients and their relatives toward PEG, and the impact of those attitudes on the decision-making process.

ELIGIBILITY:
Inclusion Criteria for patients:

* 18 years of age or older
* diagnosis of ALS
* follow-up at University Medical Centre Ljubljana, Division of Neurophysiology, every 3 months
* be able to visit the study site for in-person procedures every 3 months

Inclusion Criteria for relatives:

* at least 18 years of age

Exclusion Criteria for patients:

* co-existing illness or disorder that could influence the swallowing function independently of the ALS diagnosis
* clinically significant cognitive deterioration or dementia at enrollment, as determined by the ALS study neurologist

Exclusion criteria for relatives:

* signs of probable cognitive deterioration or dementia at enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult ALS patients able to visit the study site for in-person procedures every 3 months, and their close relatives.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale (PAS) change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  PAS is an 8-point scale used to determine swallowing safety. Levels 1 and 2 are considered safe, levels >3 indicate penetration or aspiration and are considered unsafe.
Yale Residue Severity Rating Scale (YRSRS) change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  YRSRS is a validated measure of swallowing efficiency using an image-based assessment to determine post-swallow pharyngeal residue: location and severity. It is assessed using a 5-point ordinal scale (from 1=0 % residue to 5=50 % residue).
Iowa Oral Performance Instrument (IOPI) change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  IOPI is a device which measures tongue strength (in kilopascals; kPa) and endurance (in seconds) while the participant presses the bulb with the front or the base of their tongue to the hard palate.
Mann Assessment of Swallowing Ability (MASA) change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  MASA is a standard clinical swallowing assessment protocol administered by the speech-language therapist. Total score ranges from 38-200. Lower score indicates higher impairment.
Eating Assessment Tool 10 (EAT-10) change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  EAT-10 is a validated self-administered dysphagia severity symptom survey including 10 items and a five-point scale (0=no problem to 4=sever problem). Higher total score indicates higher impairment.
Swallowing Quality of Life Questionnaire (SWAL-QoL) change | At baseline and every 3 months until PEG insertion, 3 and 6 months after PEG insertion
  SWAL-QoL is a 44-item standardised psychometric scale that measures swallowing-related QoL across 10 domains. Scores for each individual domain and a total SWAL-QoL score are calculated. Total score ranges from 0-100 (100 indicating the most favourable state).
Questionnaire on Attitudes Toward PEG Tube Feeding and Insertion Procedure change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  The questionnaire comprises 10 questions. The participants specify their level of agreement on a five-point Likert-type scale (1=strongly disagree, 5= strongly agree).

SECONDARY OUTCOMES:
ALS Functional Rating Scale-Revised (ALSFRS-R) change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  ALSFRS-R is a 12-tem ALS-specific assessment of global functioning using a five-point scale (0=not able, 4= normal ability), with 48 points representing normal function.
Functional Oral Intake Scale (FOIS) change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  FOIS is a validated 7-point scale demonstrating an individual's ability of daily oral food intake (1=no oral intake, 7=total oral intake with no restrictions).
Dysphagia Outcome and Severity Scale (DOSS) change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  DOSS is a 7-point scale that rates the functional severity of dysphagia based on objective assessment and provides information on diet recommendations, independence level and type of nutrition necessary (level 7=normal swallowing function, level 1=severe dysphagia).
BMI change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  Body mass index (in kg/m^2)
Forced Vital Capacity (FVC) change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  Standard clinical respiratory assessment of FVC (in %)
Peak Cough Flow (PCF) change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  Standard clinical respiratory assessment of PCF (in L/min)
Maximal Inspiratory Pressure (MIP) change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  Standard clinical respiratory assessment of MIP (in cmH2)
Maximal Expiratory Pressure (MEP) change | Difference between baseline and PEG insertion (usually in 6-25 months after diagnosis, maximum follow-up 30 months)
  Standard clinical respiratory assessment of MEP (in cmH2)

CONTACTS AND LOCATIONS:
Overall Officials: Blaž Koritnik, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No